CLINICAL TRIAL: NCT06790849
Title: The Impact of Chronic Consumption of ETAS® for 12 Weeks on Cognitive, Affective, and Inflammatory Outcomes: A Randomised Parallel Group Placebo-controlled Feasibility Study
Brief Title: ETASCAI Pilot Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Collaborators: Amino Up Chemicals Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Piril Hepsomali, Principle Investigator, University of Reading
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: UREC 24_39
Record Dates: First submitted 2025-01-13; First posted 2025-01-24 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-03

CONDITIONS: Cognition; Affect (Mental Function); Inflammation
Keywords: ETAS®; cognition; depression; anxiety; sleep; quality of life; inflammation; tau
MeSH Terms: conditions — Inflammation; Depression; Anxiety Disorders; Pick Disease of the Brain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active 1: ETAS® (300mg) (Experimental): Subjects will consume 300mg ETAS®/day (capsule).
  Interventions: Dietary Supplement: Active 1 ETAS®
- Active 1: ETAS® (1500mg) (Active Comparator): Subjects will consume 1500mg ETAS®/day (capsule).
  Interventions: Dietary Supplement: Active 2 ETAS®
- Placebo: Matched placebo (Placebo Comparator): Subjects will consume a matched placebo capsule.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Active 1 ETAS® — 300 mg ETAS®
  Arms: Active 1: ETAS® (300mg)
Dietary Supplement: Active 2 ETAS® — 1500mg ETAS®
  Arms: Active 1: ETAS® (1500mg)
Dietary Supplement: Placebo — Matched placebo capsule
  Arms: Placebo: Matched placebo

SUMMARY:
This pilot study aims to investigate the chronic effects of ETAS® on cognitive, affective and inflammatory outcomes in healthy adults aged 60-80 years with mild to moderate subjective cognitive complaints.

DETAILED DESCRIPTION:
This pilot study will employ a double-blind, randomised, placebo-controlled parallel design to investigate the chronic effects of 12-week-long ETAS® consumption on affective, inflammatory, metabolic, and anthropometric outcomes in healthy older adults with mild to moderate subjective cognitive complaints. Thirty participants will be randomised to Intervention 1, Intervention 2, or Placebo groups where they will be consuming capsules containing 300mg ETAS®, 1500mg ETAS®, or placebo, respectively, for 12-weeks. Outcome measures will be acquired before and after a 12-week chronic supplementation. These will include cognitive measures of overall cognitive functioning, executive function, and cognitive failures; affective measures of depression and anxiety symptomatology; quality of life, and sleep; gastrointestinal symptomatology; inflammatory measures of IFN-γ, IL-1β, IL-2, IL-4, IL-6, IL-8, IL-10, IL-12p70, IL-13, TNF-α, CRP; systolic and diastolic blood pressure, as well as height, weight, hip and waist circumference. In addition, tau from plasma will be recorded at all timepoints.

ELIGIBILITY:
Inclusion Criteria:

* Aging between 60-80 years old
* Having normal vision and hearing
* Having a body mass index between 18.5 and 30
* Having mild to moderate subjective cognitive complaints

Exclusion Criteria:

* Smoking
* Having food allergies or intolerances
* Following restrictive and/or unbalanced diets
* Changing dietary intake majorly in past month
* Being diagnosed with any psychiatric or neurologic conditions (e.g. schizophrenia, depression, dementia) including eating disorders
* Being diagnosed with any cardiometabolic diseases (including type II diabetes and cardiovascular disease), or suffering from hypertension or thrombosis related disorders or suffer from thyroid disease
* Being anaemic
* Currently taking anticoagulants, antiplatelet medication, antidepressants, proton-pump inhibitors
* Currently consuming prebiotic or probiotic supplements
* Continuous antibiotic use for > 3 days within 1 month prior to enrolment
* Continuous use of weight-loss drug for > 1 month before screening
* Having inflammatory bowel disease; coeliac disease; total colectomy or bariatric surgery; irritable bowel disease; end stage renal disease; active cancer, or treatment for any cancer, in last 3 years

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2025-02-24 (Actual); Primary Completion 2025-10-22 (Actual); Study Completion 2025-10-22 (Actual)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) score | From baseline (pre intervention) to week 12 (post intervention)
  Composite measure of global cognitive function
Inflammatory biomarker levels | From baseline (pre intervention) to week 12 (post intervention)
  IFN-γ, IL-1β, IL-2, IL-4, IL-6, IL-8, IL-10, IL-12p70, IL-13, TNF-α, CRP levels from plasma

SECONDARY OUTCOMES:
Behaviour Rating Inventory of Executive Function Score | From baseline (pre intervention) to week 12 (post intervention)
  A validated questionnaire that measures inhibition, self-monitoring, planning, task monitoring, emotional control, working memory and organisation of materials.
Cognitive Failures Questionnaire Score | From baseline (pre intervention) to week 12 (post intervention)
  A validated questionnaire that measures episodes of absent-mindedness, including slow performance on focused attention tasks.
Geriatric Depression Scale scores | From baseline (pre intervention) to week 12 (post intervention)
  A validated self-report measure of depression that includes 15-items.
Geriatric Anxiety Inventory scores | From baseline (pre intervention) to week 12 (post intervention)
  A validated self-report measure of anxiety that includes 20-items.
Pittsburgh Sleep Quality Index Scores | From baseline (pre intervention) to week 12 (post intervention)
  A validated self-report measure of sleep quality.
WHOQOL-BREF score | From baseline (pre intervention) to week 12 (post intervention)
  A validated measure of quality of life
Gastrointestinal Symptom Rating Scale Scores | From baseline (pre intervention) to week 12 (post intervention)
  A validated self-report measure of gastrointestinal symptoms that includes 15-items (combined into five symptom clusters depicting Reflux, Abdominal pain, Indigestion, Diarrhoea and Constipation)
EPIC Norfolk Food Frequency Questionnaire (FFQ) | From baseline (pre intervention) to week 12 (post intervention)
  The FFQ is a validated tool for gauging the average habitual dietary intake of micro and macronutrients of an individual in the UK. Data will be processed using the FETA software.
Blood Pressure | From baseline (pre intervention) to week 12 (post intervention)
  Systolic and diastolic blood pressure (in mmHg) will be measured.
Hip and waist circumference | From baseline (pre intervention) to week 12 (post intervention)
  Hip and waist circumference (in cm) will be measured.
Body Mass Index | From baseline (pre intervention) to week 12 (post intervention)
  Weight (in kg) and height (in m) will be combined to report Body Mass Index in kg/m^2.

OTHER OUTCOMES:
Telephone Interview for Cognitive Status-40 | Baseline (pre intervention)
  A questionnaire that assesses cognitive status. It will be used to screen participants. Only individuals who score between 6 and 20 (depicting mild to moderate subjective cognitive complaints) will be included in the study.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Reading, School of Psychology and Clinical Languages, Reading, Berkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No